CLINICAL TRIAL: NCT05444088
Title: An Open-label, Multicenter Phase Ib/II Clinical Study of SHR-8068 Combined With Adebrelimab and Bevacizumab in the Treatment of Advanced Hepatocellular Carcinoma
Brief Title: Study of SHR-8068 Combined With Adebrelimab and Bevacizumab in the Treatment of Advanced Hepatocellular Carcinoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Suzhou Suncadia Biopharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHR-8068-II-201-HCC
Record Dates: First submitted 2022-06-26; First posted 2022-07-05 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Advanced Hepatocellular Carcinoma
MeSH Terms: interventions — Bevacizumab

STUDY DESIGN:
Intervention Model Description: This study is a multicenter, open-label, dose-finding and efficacy-expansion phase Ib/II study. The phase Ib design is for dose finding and dose confirmation, using modified 3+3 design; the phase II design is for efficacy expansion through randomization.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Adebrelimab in combination with Bevacizumab (Experimental)
  Interventions: Drug: Adebrelimab; Drug: Bevacizumab
- Adebrelimab in combination with Bevacizumab and SHR-8068 RP2D1 (Experimental)
  Interventions: Drug: Adebrelimab; Drug: Bevacizumab; Drug: SHR-8068
- Adebrelimab in combination with Bevacizumab and SHR-8068 RP2D2 (Experimental)
  Interventions: Drug: Adebrelimab; Drug: Bevacizumab; Drug: SHR-8068

INTERVENTIONS:
Drug: Adebrelimab — intravenous infusion
Drug: Bevacizumab — intravenous infusion
Drug: SHR-8068 — intravenous infusion
  Arms: Adebrelimab in combination with Bevacizumab and SHR-8068 RP2D1; Adebrelimab in combination with Bevacizumab and SHR-8068 RP2D2

SUMMARY:
To evaluate the tolerability and safety of SHR-8068 in combination with Adebrelimab and Bevacizumab in subjects with advanced HCC; To evaluate the efficacy of SHR-8068 in combination with Adebrelimab and Bevacizumab in subjects with advanced HCC.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18~75 years old, both male and female;
2. Stage 1: pathologically diagnosed, incurable advanced HCC subjects who have failed standard treatment or were unwilling to accept standard treatment;
3. Stage 2: pathologically diagnosed, incurable advanced HCC subjects, who have no prior immunotherapy, no more than 1 line of previous system treatment;
4. At least one measurable lesion based on RECIST v1.1 criteria;
5. Barcelona clinic liver cancer: Stage B or C;
6. ECOG PS score: 0-1 points;
7. Child-Pugh score: ≤ 7;
8. Expected survival period ≥ 3 months;
9. Adequate organ function.

Exclusion Criteria:

1. Fibrolamellar hepatocellular carcinoma, sarcomatoid hepatocellular carcinoma or mixed cholangiocarcinoma / hepatocellular carcinoma;
2. Patients with any active, known or suspected autoimmune disorder;
3. Systemic treatment with corticosteroids or other immunosuppressants within 1 month before the first dose;
4. With known severe allergic reactions to any other monoclonal antibodies;
5. Patients with known CNS metastasis or hepatic encephalopathy;
6. Patients with liver tumor burden greater than 50% of total liver in volume, or patients who have previously undergone liver transplantation;
7. Patients with symptomatic ascites or pleural effusion requiring paracentesis and drainage, or patients who have undergone ascites or pleural effusion drainage within 2 weeks before the first dose;
8. Patients with other malignancies currently or within the past 5 years;
9. Patients with hypertension which cannot be well controlled by antihypertensives;
10. Uncontrolled cardiac diseases or symptoms;
11. Patients with other potential factors that may affect the study results.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Estimated)
Dates: Start 2022-08-02 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicity | The observation period is 21 days after the first dose
Incidence and severity of grade ≥3 drug-related adverse events and serious adverse events of the two-drug or three-drug combination | The observation period is from the time when all informed subjects signed the informed consent to the end of the safety follow-up period, up to 2 years
Objective Response Rate | At the time point of every 6 or 9 weeks, up to 2 years
  determined using RECIST v1.1 criteria, defined as best overall response (complete or partial response) across all assessment time points

SECONDARY OUTCOMES:
Disease Control Rate, determined using RECIST v1.1 criteria | At the time point of every 6 or 9 weeks, up to 2 years
Progression-Free-Survival assessed by investigator | up to 2 years]

CONTACTS AND LOCATIONS:
Locations (1):
- Anhui Provincial Hospital Ethics Commitee, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: Undecided